CLINICAL TRIAL: NCT00757094
Title: Safety and Feasibility of Fasting While Receiving Chemotherapy
Status: Completed | Type: Observational
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Ali Al-Shanqeeti, King Fahad Medical City
Other Study IDs: KFMC IRB-08-040
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Fasting; Chemotherapy; Cancer
Keywords: Fasting; Chemotherapy; Cancer
MeSH Terms: conditions — Fasting; Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- I: Patients planning to observe fasting while receiving chemotherapy during the month of Ramadan

SUMMARY:
Fasting (refraining from eating and drinking) during the day is safe while receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Established diagnosis of cancer
* Signed informed consent
* Adequate CBC and chemistry to receive chemotherapy

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fasting patients who are schedulled to receive chemotherapy during the month of Ramadan
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Safety of fasting while receiving chemotherapy | two months

SECONDARY OUTCOMES:
Effect of fasting on chemotherapy side effects | two months

CONTACTS AND LOCATIONS:
Overall Officials: Ali SM Al-Shanqeeti, MD, Principal Investigator — King Fahad Medical City
Locations (1):
- King Fahad Medical City, Riyadh, Riyadh Region, Saudi Arabia

REFERENCES:
- [Background] Raffaghello L, Lee C, Safdie FM, Wei M, Madia F, Bianchi G, Longo VD. Starvation-dependent differential stress resistance protects normal but not cancer cells against high-dose chemotherapy. Proc Natl Acad Sci U S A. 2008 Jun 17;105(24):8215-20. doi: 10.1073/pnas.0708100105. Epub 2008 Mar 31. PMID 18378900
- [Background] Weindruch R, Walford RL. Dietary restriction in mice beginning at 1 year of age: effect on life-span and spontaneous cancer incidence. Science. 1982 Mar 12;215(4538):1415-8. doi: 10.1126/science.7063854.
- [Background] Ross MH, Bras G. Lasting influence of early caloric restriction on prevalence of neoplasms in the rat. J Natl Cancer Inst. 1971 Nov;47(5):1095-113. No abstract available. PMID 4330798
- [Background] Klurfeld DM, Welch CB, Lloyd LM, Kritchevsky D. Inhibition of DMBA-induced mammary tumorigenesis by caloric restriction in rats fed high-fat diets. Int J Cancer. 1989 May 15;43(5):922-5. doi: 10.1002/ijc.2910430532. PMID 2497075
- [Background] Dirx MJ, Zeegers MP, Dagnelie PC, van den Bogaard T, van den Brandt PA. Energy restriction and the risk of spontaneous mammary tumors in mice: a meta-analysis. Int J Cancer. 2003 Sep 20;106(5):766-70. doi: 10.1002/ijc.11277. PMID 12866038